CLINICAL TRIAL: NCT04135547
Title: Venous Injection Compared To intraOsseous Injection During Resuscitation of Patients With Out-of-hospital Cardiac Arrest (The VICTOR Trial)
Brief Title: Venous Injection Compared To intraOsseous Injection During Resuscitation of Patients With Out-of-hospital Cardiac Arrest
Acronym: VICTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201904039RIND
Record Dates: First submitted 2019-10-16; First posted 2019-10-22 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Emergency Medical Service; Out-of-Hospital Cardiac Arrest; Vascular Access; Intraosseous Access; Intravenous Access
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Masking Description: The intervention (IO vs IV route) on the patients with out-of-hospital cardiac arrest can not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- intra-osseous access, IO at the humeral site (Experimental): the OHCA patients receiving IO at the humeral site by paramedics in the field
  Interventions: Device: intra-osseous access vs. intra-venous access
- intravenous access; IV at the upper limb (Active Comparator): the OHCA patients receiving IV at the upper limb by paramedics in the field
  Interventions: Device: intra-osseous access vs. intra-venous access

INTERVENTIONS:
Device: intra-osseous access vs. intra-venous access — EZ-IO®: The Arrow® Intraosseous Vascular Access System from Teleflex IV-catheter: form local qualified manufactures
  Other Names: EZ-IO® vs. IV-catheter

SUMMARY:
Overall survival of patients after out-of-hospital cardiac arrest (*OHCA*) is less than 10% worldwide and in Taiwan. Interventions provided by the emergency medical system (*EMS*) before arrival at the hospital are of paramount importance to patient outcomes after OHCA. Among those interventions, the pros-and-cons of different vascular accesses, including intraosseous (*IO*) access or intravenous (*IV*) access, remained the issue of most under debate.

The objective of this study is to determine the comparative effectiveness of IO access vs IV access in patients with OHCA by a randomized controlled trial (*RCT*) in Taipei EMS. To name in short, the investigators called it a "*VICTOR* trial" standing for "Venous Injection Compared To intraOsseous injection during Resuscitation of patients with out-of-hospital cardiac arrest".

DETAILED DESCRIPTION:
Overall survival of patients after out-of-hospital cardiac arrest (*OHCA*) is less than 10% worldwide and in Taiwan. Interventions provided by the emergency medical system (*EMS*) before hospital care is of paramount importance to patient outcomes after OHCA. Among those interventions, the pros and cons of different vascular accesses, including intraosseous (*IO*) access or intravenous (*IV*) access, recently became the focus under debate.

Theoretically, IO access provides a rapidly established way to administrate medication and fluid to patients (Reference 1) and has been adopted in many acute care societies and organizations including current resuscitation guidelines (Reference 2). However, some of the recent publications questioned the outcomes of OHCA patients receiving the IO route comparing to the IV route (References 3-5). Studies showed non-different or negative outcomes of patients receiving the IO route has been severely biased through the inherent inadequacy of retrospective design (References 3-5). The three major problems of those studies were:

1. . Time to vascular access cannot be adjusted. In many EMS, IO access was allowed only after one or two failed attempts of IV route. This led to a significant selection bias.
2. . The location of vascular access was not accurately reported. As we know, medications through upper limbs arrive at the heart sooner than the lower limbs. Many paramedics tend to insert the IO needle in tibia but to inset IV catheters in the forearm vein.
3. . Post-hoc analysis with old data over 5 to 10 years. Two of the three studies were the post-hoc analysis from the data of previous studies which was conducted from 2007 to 2010 when cardiopulmonary resuscitation quality and teamwork (i.e. important confounding factors to OHCA survival) were not that emphasized and recorded.

Hence, the investigators designed the study to determine the comparative effectiveness of IO access vs IV access in patients with OHCA by a randomized controlled trial (*RCT*) in Taipei EMS. In this 2-year research plan, we will conduct a prehospital RCT to address the following question: In adult patients with non-traumatic cause of OHCA resuscitated by emergency medical technician paramedic in the prehospital setting, will receiving IO access cause a better chance of survival to discharge, sustained recovery of spontaneous circulation, and other survival outcomes like neurologically favorable status, comparing to those who receiving IV access.

To name in short, the investigators called it a "*VICTOR* trial" standing for "Venous Injection Compared To intraOsseous injection during Resuscitation of patients with out-of-hospital cardiac arrest".

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest (OHCA) activated Taipei EMS ALS team (EMTP)
* Adult ≥ 20 years old

Exclusion Criteria:

* OHCA patients with signs of obvious death, e.g. rigor mortis
* Existing do-not-attempt-resuscitation order
* Patients with cardiac arrest en route to the hospital
* OHCA patients with successful vascular access before EMTP arrival
* OHCA patients with a canceled ambulance call or being transported to the hospital before EMTP arrival
* OHCA patients with known or suspected pregnancy
* OHCA patients with traumatic cause of cardiac arrest
* OHCA patients with known or suspected < 20 years old, or > 80 years old
* OHCA patients with contraindications to IO access or IV access

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1732 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
the rate of survival to hospital discharge | up to 1 month after the OHCA event
  OHCA patients with survival to hospital discharge

SECONDARY OUTCOMES:
the time and rate of return of spontaneous circulation (*ROSC*) | up to 1 week after the OHCA event
  the time and rate of return of spontaneous circulation (*ROSC*), prehospital ROSC
survival to admission | up to 1 week after the OHCA event
  survival to admission, or in some overcrodwed hospital, surrogated by sustained ROSC > 2hrs
favorable neurologic survival staus | up to 1 month after the OHCA event
  favorable neurologic survival staus defined by CPC 1 & 2 level (CPC: cerebral performance categlory)

OTHER OUTCOMES:
subgroups analysis | through study completion, an average of half a year
  including subgroups with different ages, sexs, witnessed status, initial presenting rhythm (shockable vs. non-shockable), bystander CPR, response intervals, time to vascular access, and time to first-dose epinephrine.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chu Chiang, PhD, Principal Investigator — Dept. of Emergency Medicine, NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petitpas F, Guenezan J, Vendeuvre T, Scepi M, Oriot D, Mimoz O. Use of intra-osseous access in adults: a systematic review. Crit Care. 2016 Apr 14;20:102. doi: 10.1186/s13054-016-1277-6. PMID 27075364
- [Background] Link MS, Berkow LC, Kudenchuk PJ, Halperin HR, Hess EP, Moitra VK, Neumar RW, O'Neil BJ, Paxton JH, Silvers SM, White RD, Yannopoulos D, Donnino MW. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S444-64. doi: 10.1161/CIR.0000000000000261. No abstract available. PMID 26472995
- [Background] Kawano T, Grunau B, Scheuermeyer FX, Gibo K, Fordyce CB, Lin S, Stenstrom R, Schlamp R, Jenneson S, Christenson J. Intraosseous Vascular Access Is Associated With Lower Survival and Neurologic Recovery Among Patients With Out-of-Hospital Cardiac Arrest. Ann Emerg Med. 2018 May;71(5):588-596. doi: 10.1016/j.annemergmed.2017.11.015. Epub 2018 Jan 6. PMID 29310869
- [Background] Feinstein BA, Stubbs BA, Rea T, Kudenchuk PJ. Intraosseous compared to intravenous drug resuscitation in out-of-hospital cardiac arrest. Resuscitation. 2017 Aug;117:91-96. doi: 10.1016/j.resuscitation.2017.06.014. Epub 2017 Jun 16. PMID 28629995
- [Background] Mody P, Brown SP, Kudenchuk PJ, Chan PS, Khera R, Ayers C, Pandey A, Kern KB, de Lemos JA, Link MS, Idris AH. Intraosseous versus intravenous access in patients with out-of-hospital cardiac arrest: Insights from the resuscitation outcomes consortium continuous chest compression trial. Resuscitation. 2019 Jan;134:69-75. doi: 10.1016/j.resuscitation.2018.10.031. Epub 2018 Nov 1. PMID 30391366
- [Derived] Ko YC, Lin HY, Huang EP, Lee AF, Hsieh MJ, Yang CW, Lee BC, Wang YC, Yang WS, Chien YC, Sun JT, Ma MH, Chiang WC. Intraosseous versus intravenous vascular access in upper extremity among adults with out-of-hospital cardiac arrest: cluster randomised clinical trial (VICTOR trial). BMJ. 2024 Jul 23;386:e079878. doi: 10.1136/bmj-2024-079878. PMID 39043416